CLINICAL TRIAL: NCT03218696
Title: A Randomized, Double-blind Study to Evaluate the Efficacy and Tolerability of a Cough Syrup Containing Specific Plant Extracts (Poliflav M.A.) and Honey Versus Placebo in Cough Due to Upper Respiratory Tract Infection
Brief Title: Comparison of a Protective Cough Syrup Against Placebo on Night Cough in Children 1-5 Years Coughing Since 1- 2 Days Due to Common Cold
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Aboca Spa Societa' Agricola (Industry)
Responsible Party: Principal Investigator, Avner Herman Cohen, Prof. Herman Avner Cohen, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COM-17-0096
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Cough; Acute Upper Respiratory Tract Infection
Keywords: cough; children; Acute Upper Respiratory Tract Infection
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Parallel randomized double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: According to a predertermined list, the two products are provided in identical bottles and cartons appropriately labelled so as to ensure respect of the randomization list as well as blinding of all study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cough Syrup for adults and children (Experimental): CE Marked (authorized) medical device acting by protecting the oropharynx, in a non-pharmacological way, to reduce cough. It contains honey, plantago lanceolata, thymus vulgaris. Dosage form: syrup Dosage: 5 ml. Duration: one night
  Interventions: Device: Cough Syrup for adults and children
- Placebo (Placebo Comparator): The placebo intervention is a similar syrup of taste and colour, with general protective components and other necessary synthetic components which may have an influence on cough, without the specific natural protective components. Dosage form: syrup. Dosage: 5 ml. Duration: one night
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cough Syrup for adults and children — The intervention product is a medical device in Europe due to its non-pharmacological mode of action, which makes the product compliant to the medical device definition. It is made of specific extracts of plants (plantago and thymus) which provide the product with protective characteristics of the oropharynx. These protective features enable the syrup to reduce the irritative cough promoting stimuli on the throat, which decrease urge to cough threshhold. In addition to these extract, honey completes the formula. The product does not contain any artificial component and no preservatives.
  Other Names: Poliflav M.A.-honey cough syrup
  Arms: Cough Syrup for adults and children
Device: Placebo — The placebo intervention is a syrup of same taste and colour without the natural protective components but with the necessary synthetic preservatives and other co-sweeteners to guarantee quality and safety. The placebo has, in fact, all the features of a cough syrup since true placebo syrup is not possible in cough. The lack of specific natural protective components is weighed against the presence of other necessary substances which may still have an effect on cough, but this effect is not envisaged to be a specific protective effect.
  Arms: Placebo

SUMMARY:
The intent of this study is to see how boys and girls aged 1-5 and coughing since 1-2 days due to common cold respond to a specific protective cough syrup taken before going to bed for one night, with respect to a similar but not specific syrup (placebo). The symptoms evaluated include especially cough frequency but also cough intensity, bother, and sleep quality of the child and parents.

DETAILED DESCRIPTION:
Cough is a life saving reflex, therefore it is important, especially in pediatrics, to calm cough spells without sedating the reflex. Looking into mechanisms for cough management different from mucolytics, or sedatives, such as protection of irritated pharynx mucosa from post nasal drip or other irritating substances is theoretically sound and shows practical interesting results. A parallel comparison of efficacy and tolerability between such protective mechanism (acting through a barrier and radical scavenging action) due to natural substances (honey, plantago lanceolata and thymus vulgaris) and placebo has been looked at specifically on the clinically critical population of children coughing since 1-2 days and not more, including very young children of one year old. The intent of this study is to use the protective syrup versus placebo in children with moderate to severe night and daily cough, measured with a validated parent questionnaire. Daily cough is assessed to better describe and select the general condition of the child however only night cough parameters due to treatment are assessed. The degree of disturbance of cough is followed immediately after one night administration on all night parameters, with special interest to frequency.

Assessment of effectiveness of the protective cough syrup as compared to placebo is considered very interesting due to the mechanism of the remedy. The study looks at the effect of the syrup/placebo on the first night in order to well focus the "first" effect of a treatment on the ascending phase of the illness, such as to reduce to a minimum any interference due to natural regression of the symptom due to illness progression.

ELIGIBILITY:
Inclusion Criteria:

1. Cough attributed to infection of the upper respiratory tract present in the child for not more than 2 days.
2. Children aged 1 year to 5 (ie: 1 day before the 6th birthday, males and females)
3. Score of at least 3 to two of the following three questions relating to the evaluation of night cough: frequency of nocturnal cough, impact on the sleep of the child and impact on the sleep of the parent,
4. Score of at least 3 to all three questions assessing "daytime" cough considering the day prior to study entry.
5. Written signed consent by a parent.

Exclusion Criteria:

* 1. Children with a diagnosis of acute: laryngotracheal bronchitis, pneumonia, asthma, sinusitis, allergic rhinitis, as well as chronic cardiac condition, or cystic fibrosis or any anatomical respiratory tract anomalies.

  2. Children who received antihistamines or any cough medicine the day prior to study entry.

  3. The administration of any steroid preparation by oral administration or inhalation on the day prior to study entry.

  4. Known sensitivity to any component of placebo or to Plantago lanceolata or Thymus vulgaris, honey or any other component of the "Poliflav M.A.-honey cough syrup".

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Night cough frequency score reduction | First and only night of treatment
  Night cough frequency is the most invasive element of distress to the child and family. The questionnaire rating night cough is filled in the morning following enrollment, relating to the passed night. The basal night score is the score of the night before enrollment.

SECONDARY OUTCOMES:
night cough intensity score reduction | First and only night of treatment
  All these other elements constitute cough invasiveness into the quality of life of child and parents
night cough bothersomeness score reduction | First and only night of treatment
  All these other elements constitute cough invasiveness into the quality of life of child and parents
reduction of influence of cough on child sleep score | First and only night of treatment
  All these other elements constitute cough invasiveness into the quality of life of child and parents
reduction of influence of cough on parent sleep score | First and only night of treatment
  All these other elements constitute cough invasiveness into the quality of life of child and parents
reduction of influence of cough on combined night score | First and only night of treatment
  All these other elements constitute cough invasiveness into the quality of life of child and parents

CONTACTS AND LOCATIONS:
Overall Officials: Herman A Cohen, Prof., Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Pediatric Community Ambulatory Clinic - Petach-Tikva, Petah Tikva
  - Pediatric Community Ambulatory Clinic, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eccles R. The powerful placebo in cough studies? Pulm Pharmacol Ther. 2002;15(3):303-8. doi: 10.1006/pupt.2002.0364. PMID 12099783
- [Background] Eccles R. Mechanisms of the placebo effect of sweet cough syrups. Respir Physiol Neurobiol. 2006 Jul 28;152(3):340-8. doi: 10.1016/j.resp.2005.10.004. Epub 2005 Dec 2. PMID 16326149
- [Background] Hurst JR, Saleh AD. Neither anti-inflammatory nor antibiotic treatment significantly shortens duration of cough in acute bronchitis compared with placebo. Evid Based Med. 2014 Jun;19(3):98. doi: 10.1136/eb-2013-101643. Epub 2014 Jan 22. No abstract available. PMID 24453088
- [Background] Dicpinigaitis PV, Colice GL, Goolsby MJ, Rogg GI, Spector SL, Winther B. Acute cough: a diagnostic and therapeutic challenge. Cough. 2009 Dec 16;5:11. doi: 10.1186/1745-9974-5-11. PMID 20015366
- [Background] Canciani M, Murgia V, Caimmi D, Anapurapu S, Licari A, Marseglia GL. Efficacy of Grintuss(R) pediatric syrup in treating cough in children: a randomized, multicenter, double blind, placebo-controlled clinical trial. Ital J Pediatr. 2014 Jun 10;40:56. doi: 10.1186/1824-7288-40-56. PMID 24917119
- [Background] Cohen HA, Rozen J, Kristal H, Laks Y, Berkovitch M, Uziel Y, Kozer E, Pomeranz A, Efrat H. Effect of honey on nocturnal cough and sleep quality: a double-blind, randomized, placebo-controlled study. Pediatrics. 2012 Sep;130(3):465-71. doi: 10.1542/peds.2011-3075. Epub 2012 Aug 6. PMID 22869830
- [Background] Cohen HA, Hoshen M, Gur S, Bahir A, Laks Y, Blau H. Efficacy and tolerability of a polysaccharide-resin-honey based cough syrup as compared to carbocysteine syrup for children with colds: a randomized, single-blinded, multicenter study. World J Pediatr. 2017 Feb;13(1):27-33. doi: 10.1007/s12519-016-0048-4. Epub 2016 Jul 15. PMID 27457790
- [Background] Paul IM. Therapeutic options for acute cough due to upper respiratory infections in children. Lung. 2012 Feb;190(1):41-4. doi: 10.1007/s00408-011-9319-y. Epub 2011 Sep 4. PMID 21892785
- [Background] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- [Background] Paul IM, Yoder KE, Crowell KR, Shaffer ML, McMillan HS, Carlson LC, Dilworth DA, Berlin CM Jr. Effect of dextromethorphan, diphenhydramine, and placebo on nocturnal cough and sleep quality for coughing children and their parents. Pediatrics. 2004 Jul;114(1):e85-90. doi: 10.1542/peds.114.1.e85. PMID 15231978
- [Background] Yoder KE, Shaffer ML, La Tournous SJ, Paul IM. Child assessment of dextromethorphan, diphenhydramine, and placebo for nocturnal cough due to upper respiratory infection. Clin Pediatr (Phila). 2006 Sep;45(7):633-40. doi: 10.1177/0009922806291014. PMID 16928841
- [Background] Dicpinigaitis PV, Bhat R, Rhoton WA, Tibb AS, Negassa A. Effect of viral upper respiratory tract infection on the urge-to-cough sensation. Respir Med. 2011 Apr;105(4):615-8. doi: 10.1016/j.rmed.2010.12.002. Epub 2010 Dec 24. PMID 21185164
- [Background] Nosalova G, Fleskova D, Jurecek L, Sadlonova V, Ray B. Herbal polysaccharides and cough reflex. Respir Physiol Neurobiol. 2013 Jun 1;187(1):47-51. doi: 10.1016/j.resp.2013.03.015. Epub 2013 Apr 15. PMID 23597834
- [Background] Dapkevicius A, van Beek TA, Lelyveld GP, van Veldhuizen A, de Groot A, Linssen JP, Venskutonis R. Isolation and structure elucidation of radical scavengers from Thymus vulgaris leaves. J Nat Prod. 2002 Jun;65(6):892-6. doi: 10.1021/np010636j. PMID 12088434
- [Background] Shadkam MN, Mozaffari-Khosravi H, Mozayan MR. A comparison of the effect of honey, dextromethorphan, and diphenhydramine on nightly cough and sleep quality in children and their parents. J Altern Complement Med. 2010 Jul;16(7):787-93. doi: 10.1089/acm.2009.0311. PMID 20618098